CLINICAL TRIAL: NCT04118530
Title: Long Term Arrhythmia Risk and Cardiovascular Events in Hematopoietic Stem Cell Transplant Survivors: Reveal Linq Cancer Registry Study
Brief Title: Long Term Arrhythmia Risk and Cardiovascular Events in Hematopoietic Stem Cell Transplant
Acronym: ARCHER
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: UPCC35420
Record Dates: First submitted 2019-10-05; First posted 2019-10-08 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Hematopoietic Stem Cell Transplant; Atrial Fibrillation; Atrial Flutter
Keywords: Atrial Fibrillation; Hematopoietic Stem Cell Transplant; Atrial Flutter
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hematopoietic Stem Cell Transplant (HSCT) Patients: - Patients with incidence of AF/AFL in the first 30 days of transplant
  Interventions: Other: HSCT Patients

INTERVENTIONS:
Other: HSCT Patients — Prospective, observational review of incidence of AF/AFL through Carelink remote monitoring and safety of implantation of device in this population of patients through review of standard of care follow up visits post HSCT implant

SUMMARY:
The purpose of this study is to better understand the following aims:

1. Aim 1: To evaluate the rate of recurrent Atrial Fibrillation (AF)/Atrial Flutter (AFL) in hematopoietic stem call transplant (HCST) patients with incident AF/AFL identified during the initial 30 days of the transplant
2. Aim 2: To evaluate incident episodes of 1) stroke/TIA; 2) other thromboembolic events (not stroke/TIA); 3) Heart failure events; 4) Ischemic heart events
3. Aim 3: To evaluate overall implantation safety in this population

DETAILED DESCRIPTION:
We propose a registry study in hematopoietic stem cell transplant (HSCT) patients with incident atrial fibrillation/atrial flutter (AF/AFL) during the initial 30 days of transplant who will be implanted with the Medtronic Reveal Linq Implantable Cardiac Monitor (ICM) within 90 days of HSCT. We will evaluate the rate of recurrent AF/AFL as well as incident episodes of major cardiovascular events and the safety of ICM implantation in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18
2. CHADS-VASc ≥ 2
3. Recovery of platelets to >50,000 within 90 days of incident atrial fibrillation (AF) diagnosis
4. Discharge from the incident stem cell transplant (SCT) hospitalization
5. Normal sinus rhythm at the time of consent

Exclusion Criteria:

1. Prior history of atrial fibrillation (AF) or atrial flutter
2. CHADS-VASc <2
3. Platelets <50,000 after 90 days post transplantation
4. Continued SCT hospitalization at 90 days
5. Inability to receive anticoagulation
6. AF or other arrhythmia at the time of consent
7. Current use of a class IC or III antiarrhythmic medication
8. Inability to provide informed consent/significant cognitive impairment
9. Expected survival less than one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with the diagnosis that requires them to undergo HSCT who develop incident AF/AFL in the first 30 days of transplant.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Recurrent AF/AFL episodes | 1 year
  Any recurrent episodes of AF/AFL lasting ≥2 minutes identified in ICM monitoring

SECONDARY OUTCOMES:
Incident Episodes of Interest | 1 year
  Incident episodes of: stroke/TIA; other thromboembolic events (not stroke/TIA); Heart failure events; ischemic heart events. Overall device implantation safety.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fradley, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Abramson Cancer Center at University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No